CLINICAL TRIAL: NCT00938652
Title: A Phase 3, Multi-Center, Open-Label, Randomized Study of Gemcitabine/Carboplatin, With or Without BSI-201, in Patients With ER-, PR-, and Her2-Negative Metastatic Breast Cancer
Brief Title: A Phase 3, Multi-Center Study of Gemcitabine/Carboplatin, With or Without BSI-201, in Patients With ER-, PR-, and Her2-Negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC11486; 20090301 (Other: BiPar); U1111-1119-8208 (Other: WHO)
Expanded Access: NCT01130259 (No longer available)
Record Dates: First submitted 2009-07-10; First posted 2009-07-14 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Breast Cancer
Keywords: triple negative breast cancer; metastatic breast cancer; Triple negative metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Gemcitabine; Carboplatin; iniparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm G/C (Active Comparator): gemcitabine/carboplatin on Days 1 and 8 of 21-day cycle(s)
  Interventions: Drug: gemcitabine/carboplatin
- Arm G/C/I (Experimental): gemcitabine/carboplatin on Days 1 and 8, plus iniparib on Days 1, 4, 8, and 11 of 21-day cycle(s)
  Interventions: Drug: gemcitabine/carboplatin; Drug: Iniparib

INTERVENTIONS:
Drug: gemcitabine/carboplatin — Gemcitabine 1000 mg/m2 intravenous infusion (30 ± 10 minutes)
  Carboplatin AUC 2 intravenous infusion (30 ± 10 minutes or 60 ± 10 minutes)
Drug: Iniparib — Body weight adjusted dose
  intravenous infusion (60 ± 10 minutes)
  Other Names: BSI-201; SAR240550
  Arms: Arm G/C/I

SUMMARY:
The goal of this study was to determine the effect on overall survival and progression free survival by adding iniparib (BSI-201/SAR240550) to the combination of gemcitabine/carboplatin in adult patients with triple negative breast cancer (estrogen receptor (ER)-negative, progesterone receptor (PR)-negative, and human epidermal growth factor receptor 2 (HER2)-negative).

Based on data generated by BiPar/Sanofi, it is concluded that iniparib does not possess characteristics typical of the poly (ADP-ribose) polymerase (PARP) inhibitor class. The exact mechanism has not yet been fully elucidated, however based on experiments on tumor cells performed in the laboratory, iniparib is a novel investigational anti-cancer agent that induces gamma-H2AX (a marker of DNA damage) in tumor cell lines, induces cell cycle arrest in the G2/M phase in tumor cell lines, and potentiates the cell cycle effects of DNA damaging modalities in tumor cell lines. Investigations into potential targets of iniparib and its metabolites are ongoing.

DETAILED DESCRIPTION:
Participants were treated for 21-day cycles until disease progression, unacceptable toxicity, or consent withdrawal. After treatment discontinuation, participants were followed until end of study or death or receipt of new anticancer therapy, whichever was first.

ELIGIBILITY:
Inclusion Criteria:

- Histologically documented breast cancer (either primary or metastatic site) that is ER-negative, PR-negative, and HER2 non-overexpressing by immunohistochemistry (0, 1) or fluorescence in situ hybridization (FISH).

Triple-negative tumors were defined by the following criteria:

* HER2-non-overexpressing: FISH-negative (defined by ratio <2.2) or, immunohistochemical (IHC) 0, IHC 1+ or, IHC 2+ or IHC 3+ and FISH-negative.
* ER- and PR-negative: <10% tumor staining by immunohistochemistry (IHC).

  * Never having received chemotherapy for metastatic disease or, having received 1 or 2 prior chemotherapy regimens in the metastatic setting (Prior adjuvant/neoadjuvant therapy was allowed);
  * Metastatic breast cancer (Stage IV) with measurable disease by RECIST 1.1 criteria;
  * Female, ≥18 years of age;
  * Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
  * Organ and marrow function as follows: absolute neutrophil count (ANC) ≥1500/mm3, platelets ≥100,000/dL, hemoglobin ≥9 g/dL, bilirubin ≤1.5 mg/dL, serum creatinine ≤1.5 mg/dL or creatinine clearance ≥60 mL/min, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 times the upper limit of normal if no liver involvement or ≤5 times the upper limit of normal with liver involvement;
  * Radiation therapy completed at least 14 days before study dosing on day 1; radiated lesions may not have served as measurable disease;
  * Central nervous system metastases allowed if subject did not require steroids, whole brain radiation therapy (XRT), gamma/cyber knife, and brain metastases were clinically stable without symptomatic progression;
  * For women of child bearing potential, documented negative pregnancy test within two weeks of study entry and agreement to acceptable birth control during the duration of the study therapy;
  * Tissue block (primary or metastatic) or readily available fresh frozen tumor tissue for PARP expression and other pharmacogenomic studies recommended (although its absence will not exclude subjects from participating);
  * No other diagnosis of malignancy (with exception of non melanoma skin cancer or a malignancy diagnosed ≥5 years ago);
  * Obtained informed consent;
  * Capability to understand and comply with the protocol and signed informed consent document.

Exclusion Criteria:

* Systemic anticancer therapy within 14 days of the first dose of study drug;
* Prior treatment with gemcitabine, carboplatin, cisplatin or iniparib
* Had not recovered to grade ≤1 from adverse events (AEs) per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v3.0 or to within 10% of baseline values due to investigational drugs or other medications administered more than 30 days prior to study enrollment;
* Major medical conditions that might have affected study participation (e.g. uncontrolled pulmonary, renal, or hepatic dysfunction, uncontrolled infection, cardiac disease);
* Concurrent radiation therapy intended to treat primary tumor not permitted throughout the course of the study; palliative radiation was acceptable;
* Leptomeningeal disease or brain metastases requiring steroids or other therapeutic intervention;
* Pregnancy or breastfeeding;
* Inability or unwillingness to abide by the study protocol or cooperate fully with the investigator or designee.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2009-07; Primary Completion 2011-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
progression free survival | until cut-off date established from deaths rate
  Progression free survival was defined as the time interval from the date of randomization to the date of first disease progression (as assessed by Independent Radiologic Review (IRR) based on Response Evaluation Criteria in Solid Tumor (RECIST) criteria), or the date of death due to any cause, whichever occurred first.
  In the absence disease progression or death, the participant was censored at the date of the last valid tumor assessment performed before the cut-off date.
Overall survival | until cut-off date established from deaths rate
  Overall survival was defined as the time interval from the date of randomization to the date of death due to any cause.
  In the absence of confirmation of death, participant was censored at the last date he/she was known to be alive, or at the cut-off date, whichever was earlier.

SECONDARY OUTCOMES:
Best overall response | until treatment discontinuation (assessment at the end of cycle 2 then every other cycle)
  Best overall response was defined as the best evaluation observed through the entire treatment period as assessed by Independent Radiologic Review [IRR] based on Response Evaluation Criteria in Solid Tumor (RECIST) criteria.
Objective response rate | until treatment discontinuation (assessment at the end of cycle 2 then every other cycle)
  Objective response rate was defined as the percentage of patients with IRR confirmed partial response or complete response prior to disease progression or treatment discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (102):
- United States (102):
  - Research Site, Birmingham, Alabama
  - Research Site, Sedona, Arizona
  - Research Site, Jonesboro, Arkansas
  - Research Site, Alhambra, California
  - Research Site, Bakersfield, California
  - Research Site, Campbell, California
  - Research Site, Fullerton, California
  - Research Site, Lancaster, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Nothridge, California
  - Research Site, Oxnard, California
  - Research Site, Palo Alto, California
  - Research Site, Pomona, California
  - Research Site, Redondo Beach, California
  - Research Site, San Francisco, California
  - Research Site, Santa Barbara, California
  - Research Site, Santa Maria, California
  - Research Site, Sylmar, California
  - Research Site, Vallejo, California
  - Research Site, Westlake Village, California
  - Research Site, Whittier, California
  - Research Site, Denver, Colorado
  - Research Site, Grand Junction, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Bonita Springs, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Ocoee, Florida
  - Research Site, Orange Park, Florida
  - Research Site, Orlando, Florida
  - Research Site, Port Saint Lucie, Florida
  - Research Site, Albany, Georgia
  - Research Site, Athens, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Overland Park, Kansas
  - Research Site, Westwood, Kansas
  - Research Site, Baltimore, Maryland
  - Research Site, Chevy Chase, Maryland
  - Research Site, Westminster, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Royal, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Jackson, Mississippi
  - Research Site, Columbia, Missouri
  - Research Site, St Louis, Missouri
  - Reserach Site, Billings, Montana
  - Research Site, Grand Island, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Hooksett, New Hampshire
  - Research Site, Morristown, New Jersey
  - Research Site, Sparta, New Jersey
  - Research Site, Santa Fe, New Mexico
  - Research Site, Amsterdam, New York
  - Research Site, East Setauket, New York
  - Research Site, New York, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Reserach Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Reserach Site, Columbia, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Bedford, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Fredericksburg, Texas
  - Research Site, Houston, Texas
  - Research Site, Tyler, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Fairfax, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Suffolk, Virginia
  - Research Site, Kennewick, Washington
  - Research Sites, Seattle, Washington
  - Research Site, Vancouver, Washington
  - Research Site, Yakima, Washington

REFERENCES:
- [Derived] O'Shaughnessy J, Schwartzberg L, Danso MA, Miller KD, Rugo HS, Neubauer M, Robert N, Hellerstedt B, Saleh M, Richards P, Specht JM, Yardley DA, Carlson RW, Finn RS, Charpentier E, Garcia-Ribas I, Winer EP. Phase III study of iniparib plus gemcitabine and carboplatin versus gemcitabine and carboplatin in patients with metastatic triple-negative breast cancer. J Clin Oncol. 2014 Dec 1;32(34):3840-7. doi: 10.1200/JCO.2014.55.2984. Epub 2014 Oct 27. PMID 25349301